CLINICAL TRIAL: NCT06565832
Title: Reproducibility of Virtual Exercise Assessments Versus Face-to-face Exercise Testing in Adults With Cystic Fibrosis - a Pilot Feasibility Study
Brief Title: Reproducibility of Virtual Exercise Assessments Versus Face-to-face Exercise Testing in Adults With Cystic Fibrosis
Acronym: RExA-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RExA-CF V3
Record Dates: First submitted 2024-08-14; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Cystic Fibrosis
Keywords: Exercise testing
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual exercise testing via video link (Active Comparator): The One-Minute Sit-to-Stand test and the Chester Step test will be completed via a video link call with the participant and the research team.
  Interventions: Procedure: One-Minute Sit-to-Stand Test; Procedure: Chester Step Test
- Face-to-Face exercise testing (Active Comparator): The One-Minute Sit-to-Stand test and the Chester Step test will be completed face to face at a hospital appointment with the participant and the research team.
  Interventions: Procedure: One-Minute Sit-to-Stand Test; Procedure: Chester Step Test

INTERVENTIONS:
Procedure: One-Minute Sit-to-Stand Test — This test involves sitting down and standing up from a normal height chair (can be a dining room or kitchen chair at home) for one minute. Participants can rest or stop at any time if fatigued. Participants will be asked to record your heart rate and oxygen levels before and after the test and will be given a monitor to do this with if they do not already have one. This test should take a maximum of 5 minutes.
Procedure: Chester Step Test — This test involves the participant stepping up and down off of a step (this can be a bottom stair or doorstep at home) keeping up with the beat of a recording. The speed of the beat increases every 2 minutes, and the test continues until the participant cannot keep up with the pace, wish to stop or the test ends which takes 10 minutes. Participants will be asked to record heart rate and oxygen levels before and after the test. This test should take a maximum of 15 minutes.

SUMMARY:
RExA-CF is investing if results from exercise tests (the Chester Step Test and the One-Minute Sit-to-Stand test) completed face to face are comparable to results of the same tests completed via a virtual teleconferencing platform. The study involves two exercise testing sessions (one face-to-face and one via a video link), with participants being randomised to complete the two exercise tests (the 1-minute sit-to-stand test and the Chester Step test). The two testing sessions will be completed within three weeks of each other, the order of which will be randomly allocated. One session will be completed face-to-face during a pre-arranged visit to the hospital, the other test session will be completed through a video call at a time convenient to the participants. After the second testing session participants will be asked some questions about the face-to-face and video tests to get their views about the two formats.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis (as confirmed by standard criteria)
* Sixteen years of age or over
* Home internet access
* Stable CF disease as judged by the medical team
* Registered with the Royal Brompton Hospital adult CF team

Exclusion Criteria:

* Inability to give consent for treatment or measurement
* Current participation in another interventional study
* Current moderate haemoptysis (greater than streaking in the sputum)
* Pregnancy
* Forced expiratory volume in 1 second (FEV1) below 30% predicted
* Dependency upon oxygen therapy (with home oxygen concentrators or portable oxygen cylinders) or non-invasive ventilation (NIV)
* Current neurological or musculoskeletal injury which would prevent completion of exercise tests
* Inability to complete the second set of exercise tests within three weeks

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Aerobic Capacity from the Chester Step test | Completed at week 0 and within 2 weeks of first test
  This test involves the participant stepping up and down off of a step (this can be a bottom stair or doorstep at home) keeping up with the beat of a recording. The speed of the beat increases every 2 minutes, and the test continues until the participant cannot keep up with the pace, wish to stop or the test ends which takes 10 minutes. Participants will be asked to take their heart rate and oxygen levels before and after the test using a provided pulse-oximeter. This test should take a maximum of 15 minutes. The results of the test will be used to calculate the participants aerobic capacity (range 0-60)
Number of sit to stands completed during One-Minute Sit-to-Stand test | Completed at week 0 and within 2 weeks of first test
  This test involves the participant sitting down and standing up from a normal height chair (can be a dining room or kitchen chair at home) for one minute. Participants can rest or stop at any time if fatigued. This test should take a maximum of 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma E Stanford, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, Guy's and St Thomas's NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No